CLINICAL TRIAL: NCT04869124
Title: Effects of Dapagliflozin on Blood Volume Status and Vascular Function in Clinically Compensated Heart Failure Patients After an Acute Heart Failure Event.
Brief Title: Dapagliflozin on Volume Vascular Outcomes.
Acronym: DAPA-VOLVO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Frank Ruschitzka (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Frank Ruschitzka, Prof. Dr. med., University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESR-20-20601; 2020-004143-89 (EudraCT Number)
Record Dates: First submitted 2021-01-04; First posted 2021-05-03 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure，Congestive
Keywords: heart failure; congestive; hospitalization; blood volume; vascular function
MeSH Terms: conditions — Heart Failure | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: A double-blind randomized placebo-controlled phase IV clinical trial.
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Active Comparator): Dapagliflozin tablet (10mg/tablet), orally, once daily for 12 weeks.
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Placebo tablet, matching Dapglilflozin, orally, once daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin propanediol (FORXIGA) tablet: 10 mg once daily p.o. on top of recommended standard therapy, duration of administration: 12 weeks.
  Other Names: Forxiga
  Arms: Dapagliflozin
Drug: Placebo — Placebo tablet, matching Dapagliflozin, once daily p.o. on top of recommended standard therapy, duration of administration: 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of the DAPA-VOLVO trial is to investigate the effects of Dapagliflozin on top of recommended standard therapy on volume status and vascular function in clinically stable de novo or chronic heart failure patients after hospitalization because of an acute decompensated heart failure event.

DETAILED DESCRIPTION:
Recent clinical trials found that Dapagliflozin can reduce the risk of cardiovascular events, hospitalization and death in heart failure (HF) patients with reduced left ventricular ejection fraction (HFrEF) in the presence of absence of diabetes. Additional trials are ongoing to investigate whether these results can be translated also to HF-patients with preserved ejection fraction (HFpEF). However, the underlying mechanisms leading to the improved clinical outcomes are not completely understood but the beneficial effects of Dapagliflozin on volume status and vascular function are discussed as potential key factors. This study is designed as a mechanistic study to investigate the impact of Dapagliflozin on volume status and vascular function in clinically stable de novo or chronic heart failure patients after hospitalization/ ambulatory care because of an acute decompensated heart failure (ADHF) event. After being informed about the study and potential risks all patients given written informed consent will be screened for the defined eligibility criteria and thereafter randomized in a double-blind manner (patients, investigators) 1:1 ratio to either receive the sodium-glucose co-transporter 2 inhibitor (SGLT2i) Dapagliflozin (10mg/day) or Placebo on top of recommended standard therapy for in total 12 weeks. The results of this study may provide new mechanistic insight into the beneficial effects of Dapagliflozin on volume regulation and vascular function and have great potential to contribute to change current clinical guidelines in the management of patients with heart failure.

ELIGIBILITY:
Inclusion criteria:

1. Male or female, age of 18 or older;
2. Patients with documented diagnosis of chronic or de novo heart failure (NYHA II-IV) and clinically stabilized (considered for hospital discharge) after hospitalization/ ambulatory care because of an acute decompensated (congestive) heart failure (ADHF) event;
3. eGFR ≥ 30 mL/min/1.73 m2 (CKD-EPI formula) at enrolment;
4. Provision of signed informed consent prior to any study specific procedure;

Exclusion criteria:

1. Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product;
2. Receiving therapy with an SGLT2 inhibitor within 8 weeks prior to enrolment or previous intolerance of an SGLT2 inhibitor;
3. Participation in another study with investigational drug within the 30 days preceding and during the present study;
4. Type 1 diabetes mellitus;
5. Symptomatic hypotension or systolic blood pressure <90 mmHg at 2 out of 3 measurements either at visit 1 or visit 2;
6. Coronary revascularization (percutaneous coronary intervention because of STEMI or coronary artery bypass grafting) or valvular repair/replacement within 12 weeks prior to enrolment or planned to undergo any of these operations after randomization;
7. Implantation of a CRT device within 12 weeks prior to enrolment or intent to implant a CRT device during 12 weeks of study observation period if indicated according to the actual guidelines [11];
8. Previous cardiac transplantation or implantation of a ventricular assistance device or similar device, or implantation expected after randomization;
9. HF due to restrictive cardiomyopathy, active myocarditis, constrictive pericarditis, hypertrophic obstructive cardiomyopathy or uncorrected primary valvular disease;
10. Symptomatic bradycardia or second or third degree heart block without a pacemaker;
11. Severe (eGFR <20 mL/min/1.73 m2 by CKD-EPI), unstable or rapidly progressing renal disease;
12. Women who are pregnant or breast feeding;
13. Intention to become pregnant during the course of the study;
14. Known or suspected non-compliance, drug or alcohol abuse;
15. Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant;
16. Patients with severely restricted liver function;
17. Patients with recurrent mycotic genital infections;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Change in relative plasma volume status (PVS). | Change between baseline (0 weeks) and after 2, 6 and 12 weeks of treatment.
  Change in relative plasma volume status (PVS) from baseline to 12 weeks of dapagliflozin treatment in comparison to placebo will be assessed. The plasma volume (PV) will be measured via optimized CO-rebreathing technique.

SECONDARY OUTCOMES:
Change in blood volume (BV). | Change between baseline (0 weeks) and after 2, 6 and 12 weeks of treatment.
  Change in BV from baseline to 12 weeks of dapagliflozin treatment in comparison to placebo will be assessed. The BV will be measured via optimized CO-rebreathing technique.
Change in red blood cell volume (RBCV). | Change between baseline (0 weeks) and after 2, 6 and 12 weeks of treatment.
  Change in RBCV from baseline to 12 weeks of dapagliflozin treatment in comparison to placebo will be assessed. The RBCV will be measured via optimized CO-rebreathing technique.
Change in total hemoglobin mass (Hbmass). | Change between baseline (0 weeks) and after 2, 6 and 12 weeks of treatment.
  Change in Hbmass from baseline to 12 weeks of dapagliflozin treatment in comparison to placebo will be assessed. The Hbmass will be measured via optimized CO-rebreathing technique.
Change in extracellular to total body water ratio (ECW/TBW). | Change between baseline (0 weeks) and after 2, 6 and 12 weeks of treatment.
  Change in ECW/TBW ratio from baseline to 12 weeks of dapagliflozin treatment in comparison to placebo will be assessed. The ECW/TBW ratio will be measured via direct segmental multi-frequency bioelectrical impedance analaysis (DSM-BIA).
Change in intracellular to total body water ratio (ICW/TBW). | Change between baseline (0 weeks) and after 2, 6 and 12 weeks of treatment.
  Change in ICW/TBW ratio from baseline to 12 weeks of dapagliflozin treatment in comparison to placebo will be assessed. The ICW/TBW ratio will be measured via direct segmental multi-frequency bioelectrical impedance analaysis (DSM-BIA).
Change in flicker-light induced retinal arteriolar dilatation (FIDa). | Change between baseline (0 weeks) and after 12 weeks of treatment.
  Change in FIDa from baseline to 12 weeks of dapagliflozin treatment in comparison to placebo will be assessed. The FIDa will be measured via dynamic retinal vessel analysis (DVA).
Change in flicker-light induced retinal venular dilatation (FIDv). | Change between baseline (0 weeks) and after 12 weeks of treatment.
  Change in FIDv from baseline to 12 weeks of dapagliflozin treatment in comparison to placebo will be assessed. The FIDv will be measured via dynamic retinal vessel analysis (DVA).
Change in retinal arterial to venous ratio (AVR). | Change between baseline (0 weeks) and after 12 weeks of treatment.
  Change in AVR from baseline to 12 weeks of dapagliflozin treatment in comparison to placebo will be assessed. The AVR will be measured via static retinal vessel analysis (SVA).
Change in pulse wave velocity (PWV). | Change between baseline (0 weeks) and after 12 weeks of treatment.
  Change in PWV from baseline to 12 weeks of dapagliflozin treatment in comparison to placebo will be assessed. The PWV as measure of arterial stiffness (AS) will be assessed via planar tonometry pulse wave analysis (PWA).
Change in flow-mediated dilatation (FMD) of the brachial artery. | Change between baseline (0 weeks) and after 12 weeks of treatment.
  Change in FMD from baseline to 12 weeks of dapagliflozin treatment in comparison to placebo will be assessed. The FMD as measure of endothelial function will be assessed via arm sonography and short-term cuff-mediated arm ischemia.
Change in glyceryl-trinitrate-(GTN) induced dilatation of the brachial artery. | Change between baseline (0 weeks) and after 12 weeks of treatment.
  Change in GTN-induced dilatation of the brachial artery from baseline to 12 weeks of dapagliflozin treatment in comparison to placebo will be assessed. The GTN-induced dilatation of the brachial artery will be measured via arm sonography and sublingual GTN-puff.

OTHER OUTCOMES:
First episode of worsening of heart failure (WHF). | From baseline (0 weeks) to 12 weeks of treatment.
  The first episode of WHF from baseline to 12 weeks of dapagliflozin treatment in comparison to placebo will be assessed. WHF is defined as requiring intensification of therapy in the ambulatory or hospital setting including i.v. diuretics, i.v. nitrates, or other medications for HF, or institution of mechanical or ventilator support.
Change in Kansas City cardiomyopathy questionnaire (KCCQ) score. | Change between baseline (0 weeks) and after 12 weeks of treatment.
  Change in KCCQ overall score from baseline to 12 weeks of dapagliflozin treatment in comparison to placebo will be assessed. The KCCQ as a measure of HF-related quality of life will be assessed as self-administered 23-itmes questionnaire.
  The KCCQ-score range: from 0 (worst) to 100 (best).
Change in Pittsburgh sleep quality index (PSQI) score. | Change between baseline (0 weeks) and after 12 weeks of treatment.
  Change in PSQI total score from baseline to 12 weeks of dapagliflozin treatment in comparison to placebo will be assessed.The PSQI as a measure of sleep quality will be assessed as self-administered 19-itmes questionnaire.
  The PSQI-score range: 0 (best) to 21 (worst).
Change in left ventricular ejection fraction (LVEF). | Change between baseline (0 weeks) and after 12 weeks of treatment.
  Change LVEF from baseline to 12 weeks of dapagliflozin treatment in comparison to placebo will be assessed. The LVEF will be measured via transthoracic echocardiography (TTE).
Change in pulmonary artery systolic pressure (PASP). | Change between baseline (0 weeks) and after 12 weeks of treatment.
  Change PASP from baseline to 12 weeks of dapagliflozin treatment in comparison to placebo will be assessed. The PASP will be measured via transthoracic echocardiography (TTE).
Change in peak oxygen uptake (VO2peak). | Change between baseline (0 weeks) and after 12 weeks of treatment.
  Change in VO2peak from baseline to 12 weeks of dapagliflozin treatment in comparison to placebo will be assessed. The VO2peak as a measure of aerobic capacity will be assessed via cardio-pulmonary exercise test (CPET).
Change in ventilation to end-tidal carbon dioxide partial pressure (VE/ETCO2) slope. | Change between baseline (0 weeks) and after 12 weeks of treatment.
  Change in VE/PETCO2 slope from baseline to 12 weeks of dapagliflozin treatment in comparison to placebo will be assessed. The VE/PETCO2 slope as a prognostic marker in HF will be assessed via cardio-pulmonary exercise test (CPET).
Change in stimulus response to cold pressor test (CPT) of muscle sympathetic nerve activity (MSNA) . | Change between baseline (0 weeks) and after 12 weeks of treatment.
  Change in MSNA stimulus response from baseline to 12 weeks of dapagliflozin treatment in comparison to placebo will be assessed. The MSNA will be measured via transcutanous microneurography before and after cold pressor test (CPT).
Change in leg skin tissue sodium content (Skin-Na). | Change between baseline (0 weeks) and after 12 weeks of treatment.
  Change in Skin-Na from baseline to 12 weeks of dapagliflozin treatment in comparison to placebo will be assessed. The Skin-Na will be measured via 23Na-magnetic resonance imaging (23Na-MRI) technique.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Ruschitzka, M.D., Principal Investigator — Cardiology, University Heart Center Zurich
Locations (1):
- University Heart Center Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bitos K, Laptseva N, Haider T, Rossi VA, Nagele MP, Barthelmes J, Ruschitzka F, Sudano I, Flammer AJ. Effects of dapagliflozin on blood volume status and vascular outcomes in clinically stabilized heart failure patients after an acute decompensated heart failure event (DAPA-VOLVO study): Protocol of a double-blind randomized controlled clinical trial. PLoS One. 2025 Jul 2;20(7):e0325668. doi: 10.1371/journal.pone.0325668. eCollection 2025. PMID 40601599